CLINICAL TRIAL: NCT01759576
Title: An Open-Label, Single-Dose Study to Evaluate JNJ-28431754 Pharmacokinetics, Pharmacodynamics and Safety in Non-Diabetic Subjects With Varying Degrees of Renal Function
Brief Title: A Study to Assess the Pharmacokinetics, Pharmacodynamics, and Safety of Canagliflozin (JNJ-28431754) in Volunteers With Varying Degrees of Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014761; 28431754DIA1003 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2012-12-24; First posted 2013-01-03 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Renal Insufficiency; Healthy
Keywords: Renal Insufficiency; Healthy; Canagliflozin (JNJ-28431754); Pharmacokinetics; Pharmacodynamics; Dialysis
MeSH Terms: conditions — Renal Insufficiency | interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (normal kidney function) (Experimental): Each volunteer will receive a single dose of canagliflozin (JNJ-28431754) on Day 1
  Interventions: Drug: Canagliflozin (JNJ-28431754)
- Group 2 (mild kidney impairment) (Experimental): Each volunteer will receive a single dose of canagliflozin (JNJ-28431754) on Day 1
  Interventions: Drug: Canagliflozin (JNJ-28431754)
- Group 3 (moderate kidney impairment) (Experimental): Each volunteer will receive a single dose of canagliflozin (JNJ-28431754) on Day 1
  Interventions: Drug: Canagliflozin (JNJ-28431754)
- Group 4 (severe kidney impairment) (Experimental): Each volunteer will receive a single dose of canagliflozin (JNJ-28431754) on Day 1
  Interventions: Drug: Canagliflozin (JNJ-28431754)
- Group 5 (hemodialysis) (Experimental): Each volunteer will receive a single dose of canagliflozin (JNJ-28431754) on Day 1 following completion of hemodialysis. Approximately 10 days later, each volunteer will receive another single dose of canagliflozin before hemodialysis begins.
  Interventions: Drug: Canagliflozin (JNJ-28431754)

INTERVENTIONS:
Drug: Canagliflozin (JNJ-28431754) — Volunteers in groups 1 through 4 will receive one 200mg tablet orally (by mouth) on Day 1. Volunteers in group 5 will receive one 200mg tablet orally on Day 1 (one hour after hemodialysis) followed, approximately 10 days later, by one 200mg tablet orally (2 hours before hemodialysis).
  Other Names: JNJ-28431754

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (ie, how the body affects the drug) and pharmacodynamics (ie, how the drug affects the body) of canagliflozin (JNJ-28431754) after administration of a single dose to non-diabetic volunteers with normal kidney function and non-diabetic volunteers with varying degrees of kidney impairment (including volunteers with end-stage renal disease requiring hemodialysis).

DETAILED DESCRIPTION:
This study will be an open label (all volunteers and study staff know the identity of the assigned treatment), single-dose, multicenter (the study will be conducted at more than one center), parallel-group study (each group of volunteers will be treated at the same time) to assess the pharmacokinetics and pharmacodynamics of canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus) in volunteers with varying degrees of kidney function. The study will consist of 3 phases: a screening phase, an open-label treatment phase, and an end-of study (or follow-up) phase. Volunteers will be assigned to 1 of 5 groups (depending on kidney function): group 1 will have normal kidney function; group 2 will have mild kidney impairment; group 3 will have moderate kidney impairment; group 4 will have severe kidney impairment; and group 5 will comprise volunteers requiring hemodialysis. Volunteers in groups 1 through 4 will receive a single dose of canagliflozin on Day 1. Volunteers in group 5 will receive a single dose of canagliflozin following dialysis and then, approximately 10 days later, they will receive a second dose before dialysis. Volunteers in groups 1 through 4 will participate in the study for 27 days. Volunteers in group 5 will participate in the study for 40 days.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have a body mass index (BMI = weight in kg/height in m2) between 20 and 40 kg/m2 (inclusive), and body weight not less than 50 kg
* Volunteers must smoke no more than 10 cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months before first study drug administration

Exclusion Criteria:

* History of or currently active illness considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the patient from the study or that could interfere with the interpretation of the study results
* Volunteers with end stage renal disease receiving dialysis treatment other than intermittent hemodialysis
* Volunteers with end stage renal disease who have received a renal transplantation within 1 year before screening
* Volunteers with end stage renal disease diagnosed with renal carcinoma within 1 year before screening
* Volunteers with end stage renal disease receiving immunosuppressive medications, including steroids

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin (JNJ-28431754) in varying degrees of kidney function | Up to Day 6
  Plasma concentrations of canagliflozin (JNJ-28431754) following the administration of a single dose of canagliflozin will be used to determine pharmacokinetic parameters for canagliflozin (measurements describing how the body affects the drug) in varying degrees of kidney function.
Change from baseline in 24-hour urine glucose excretion in varying degrees of kidney function | Day -1 (Baseline) to Day 3
  Change from baseline in 24-hour urine glucose excretion following the administration of a single dose of canagliflozin (JNJ-28431754) will be used to evaluate the pharmacodynamics of canagliflozin (ie, how the drug affects the body) in varying degrees of kidney function.
Plasma concentrations of canagliflozin (JNJ-28431754) metabolites in varying degrees of kidney function | Up to Day 6
  Plasma concentrations of canagliflozin (JNJ-28431754) metabolites following the administration of a single dose of canagliflozin will be used to determine pharmacokinetic parameters for canagliflozin metabolites (measurements describing how the body affects the metabolites) in varying degrees of kidney function.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (3):
- United States (3):
  - Orlando, Florida
  - Minneapolis, Minnesota
  - Knoxville, Tennessee

REFERENCES:
- [Derived] Devineni D, Curtin CR, Marbury TC, Smith W, Vaccaro N, Wexler D, Vandebosch A, Rusch S, Stieltjes H, Wajs E. Effect of hepatic or renal impairment on the pharmacokinetics of canagliflozin, a sodium glucose co-transporter 2 inhibitor. Clin Ther. 2015 Mar 1;37(3):610-628.e4. doi: 10.1016/j.clinthera.2014.12.013. Epub 2015 Feb 3. PMID 25659911
- See also: An Open-Label, Single-Dose Study to Evaluate JNJ-28431754 Pharmacokinetics, Pharmacodynamics and Safety in Non-Diabetic Subjects With Varying Degrees of Renal Function — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2175&filename=CR014761_CSR.pdf